CLINICAL TRIAL: NCT00915421
Title: Pre-Hospital Cooling in Cardiac Arrest Patients - Feasibility Pilot Study
Brief Title: Pre-Hospital Cooling in Cardiac Arrest Patients
Acronym: PRE-COOL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Emergency Medical Service of the Central Bohemian Region, Czech Republic (Other)
Collaborators: University Hospital Hradec Kralove (Other)
Responsible Party: Roman Škulec, Emergency Medical Service of the Central Bohemian Region, Czech Republic
Other Study IDs: SCK-KVK-001
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2009-06-08 (Estimated); Status verified 2009-06

CONDITIONS: Cardiac Arrest
Keywords: cardiac arrest; therapeutic hypothermia; Postresuscitative disease
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Prehospital hypothermia group: All patients included to the study
  Interventions: Procedure: Induction of therapeutic mild hypothermia

INTERVENTIONS:
Procedure: Induction of therapeutic mild hypothermia — Rapid administration of 4°C cold normal saline to the peripheral vein, dose 5 - 30 ml/kg, to decrease body core temperature below 34°C

SUMMARY:
Type of study: Pilot prospective nonrandomized feasibility clinical study.

Aim of the study: To assess the feasibility of pre-hospital therapeutic mild hypothermia in patients successfully resuscitated from out-of-hospital cardiac arrest in the setting of prehospital and hospital care in Czech republic.

Evaluated hypothesis: Pre-hospital initiation of therapeutic mild hypothermia by rapid administration of intravenous bolus of cold crystalloids is simple, safe, effective and is a feasible procedure to significantly decrease body core temperature during patient's transport to the hospital in Czech republic.

The study is observational and does not evaluate any new drug, therapeutic procedure or diagnostic procedure. It is evaluating a known therapeutic procedure, therapeutic mild hypothermia, induced by known technique, cold crystalloid infusion, widely accepted in hospital-related postresuscitative care. However, even its prehospital usage has been published.

ELIGIBILITY:
Inclusion Criteria:

* patients resuscitated from out-of-hospital cardiac arrest
* remaining comatose and requiring mechanical ventilation

Exclusion Criteria:

* cardiac arrest of traumatic etiology
* patient conscious after short cardiopulmonary resuscitation
* coma of other origin than cardiac arrest (e.g., epileptic paroxysm, intoxication etc.)
* severe acute heart failure
* accidental hypothermia below 30°C
* bradycardia requiring transcutaneous cardiac pacing
* status Do Not Resuscitate or Do Not Intubate
* severe circulatory shock
* severe life threatening cardiac arrhythmias
* severe and life threatening bleeding
* severe sepsis
* any common opinion of intervening team of unfitness of induction of therapeutic mild hypothermia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Out-of-hospital cardiac arrest patients
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-07; Primary Completion 2009-07 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Effectivity measure - reached cooling rate calculated in °C/30 min | Assessed during prehospital phase

SECONDARY OUTCOMES:
Appearance of adverse events and complications during prehospital induction of therapeutic mild hypothermia | Assessed during prehospital phase
Achievement of favourable neurological outcome at the hospital discharge | Assessed during prehospital and in-hospital phase
Overall prehospital and in-hospital mortality | Assessed during prehospital and in-hospital phase
The best neurological outcome achieved anytime during hospital stay | Assessed during in-hospital phase

CONTACTS AND LOCATIONS:
Overall Officials: Roman Skulec, MD, Principal Investigator — Emergency Medical Service of the Central Bohemian Region, Czech Republic
Locations (2):
- Czechia (2):
  - Emergency Medical Service of the Central Bohemian Region, Beroun, Central Bohemia
  - Hradec Kralove Region Emergency Medical Services, Czech republic, Hradec Králové, Region of Hradec Kralove

REFERENCES:
- [Derived] Skulec R, Truhlar A, Seblova J, Dostal P, Cerny V. Pre-hospital cooling of patients following cardiac arrest is effective using even low volumes of cold saline. Crit Care. 2010;14(6):R231. doi: 10.1186/cc9386. Epub 2010 Dec 22. PMID 21176218
- See also: Web pages of Emergency Medical Service of the Central Bohemian Region, Czech republic — http://www.uszssk.cz
- See also: Web pages of Hradec Kralove Region Emergency Medical Services, Czech republic — http://www.zzskhk.cz